CLINICAL TRIAL: NCT04817358
Title: Genetic Influences on Dental Maturation: A Twin Study
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Esra Oz, Principal Investigator, Suleyman Demirel University
Other Study IDs: 2018/232
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Dental Age Estimation Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Demirjian method: According to the Demirjian method, the development of the seven left mandibular permanent teeth (except the third molar) were rated on the eight-stage scale from A to H. Each stage of mineralization was given a score, total dental maturity score was evaluated according to standard tables for boys and girls
- Willems method: Willems' method was determined using the Demirjian calcification stages but scores were evaluated according to Willems' specific tables
- Nolla method: In the Nolla method, the development of seven left mandibular and maxillar teeth were defined on 10 stages. If the tooth was between stages an appropriate fraction (0.2, 0.5 or 0.7) was added. The total score was determined according to the tables prepared for girls and boys as recommended by Nolla

SUMMARY:
The genetics has been shown as one of the most important factor influencing the growth and development of the dentofacial complex. Dental development, one of the most reliable indicators of chronological age (CA), has been believed to be fundamentally influenced by genetics rather than environmental factors. As twins share genetic variation (100% for monozygotic and 50% for dizygotic twins) and were subjected to the similar environmental factors, the twin studies have been presented useful and effective method to researchers for investigating the influence of heredity on dental development and observing the similarities and differences among twin pairs.

Evaluation of dental development is among the most commonly used and reliable method for dental age determination using the morphological parameters of teeth on dental radiographs. Dental maturity, defined as a dental age (DA), is very important in forensic anthropology to identify cases and in dentistry for planning pedodontic and orthodontic treatment, and also determining a child's growth and developmental status.

There are many dental age estimation methods which are mostly based on the morphological evaluation of dental growth observed from dental radiographs in children In order to estimate dental age, Demirjian's, Willems' and Nolla's methods were used. All panoramic radiographs were scored by one observer to eliminate the inter-observer error.

ELIGIBILITY:
Inclusion Criteria:

* good quality of panoramic radiographs, presence of all permanent mandibular and maxillar teeth except the third molars
* healthy children with normal eruption of teeth,
* children with similiar etnic origin and socio-economic status

Exclusion Criteria:

* Children with any syndromes, congenital or developmental anomalies and systemic diseases,
* Children undergoing or with previous orthodontic treatment history,
* Children with tooth agenesis, dental trauma history

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of MZ and DZ pairs between the ages of 5.0 and 12.9 who attended to the Department of Pedodontics at Suleyman Demirel University and underwent radiological examination for any dental reason during the dental treatment period from January 2018 to January 2021
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Demirjian method | up to 3 years
  the development of the seven left mandibular permanent teeth (except the third molar) were rated on the eight-stage scale from A to H. Each stage of mineralization was given a score, total dental maturity score was evaluated according to standard tables for boys and girls

SECONDARY OUTCOMES:
Willems method | up to 3 years
  Willems' method was determined using the Demirjian calcification stages but scores were evaluated according to Willems' specific tables

OTHER OUTCOMES:
Nolla method | up to 3 years
  In the Nolla method, the development of seven left mandibular and maxillar teeth were defined on 10 stages. If the tooth was between stages an appropriate fraction (0.2, 0.5 or 0.7) was added. The total score was determined according to the tables prepared for girls and boys as recommended by Nolla

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University Faculty of Dentistry, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided